CLINICAL TRIAL: NCT03153657
Title: Preemptive Use of Piroxicam-beta-Cyclodextrin on Tooth Sensitivity Caused by In-office Bleaching: Randomized, Triple-blind, Controlled Clinical Trial
Brief Title: Piroxicam-beta-Cyclodextrin on Tooth Sensitivity Caused by In-office Bleaching
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, Aline Carvalho Peixoto, Principal Investigator, Universidade Federal de Sergipe
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Univ Federal de Sergipe
Record Dates: First submitted 2017-04-14; First posted 2017-05-15 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-05

CONDITIONS: Tooth Sensitivity; Toothache
Keywords: Tooth Bleaching
MeSH Terms: conditions — Dentin Sensitivity; Toothache | interventions — piroxicam-beta-cyclodextrin; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple Blind (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Piroxicam-beta-Cyclodextrin (Experimental): Intervention: Drug Piroxicam-beta-Cyclodextrin
  Interventions: Drug: Piroxicam-Beta-Cyclodextrin; Drug: Placebo
- Placebo (Placebo Comparator): Intervention: Drug Placebo
  Interventions: Drug: Piroxicam-Beta-Cyclodextrin; Drug: Placebo

INTERVENTIONS:
Drug: Piroxicam-Beta-Cyclodextrin — The patients will receive a single-dose of Piroxicam-Beta-Cyclodextrin (20 mg) thirty minutes before the bleaching procedure.
  Other Names: Cycladol (20mg) capsule
Drug: Placebo — The patients will receive a single-dose of placebo with the same presentation of the experimental drug thirty minutes before the bleaching procedure.
  Other Names: Starch capsule made to mimic Piroxicam-Beta-Cyclodextrin

SUMMARY:
Objectives: This study aims to evaluate the effectiveness of preemptive administration of non-steroidal anti-inflammatory Piroxicam-beta-Cyclodextrin on risk and level of tooth sensitivity caused by in-office bleaching procedures using 35% hydrogen peroxide.

Fifty patients will be selected for this triple-blind, randomized, cross-over, placebo-controlled clinical trial. Piroxicam-beta-Cyclodextrin (200 mg) or placebo will be administrated in a single-dose thirty minutes prior to bleaching procedure. The whitening treatment with 35% hydrogen peroxide will be carried out in two sessions with a 7-day interval. Tooth sensitivity will be assessed Immediately before bleaching agent removal and up to 24 hours after each session the procedure using analog visual and verbal scales. Color alteration will be assessed by a bleach guide scale 7 days after each session. Relative risk to sensitivity will be calculated and adjusted by session; while comparison of overall risk will performed by Fisher's exact test. Data on the sensitivity level for both scales and color shade will be subjected to the Mann-Whitney and Friedman tests, respectively (α = 0.05).

DETAILED DESCRIPTION:
Methods & Materials:

This clinical trial was approved by the Scientific Review Committee and by the Ethics Committee on Research Involving Humans at the University Hospital of the Federal University of Sergipe (CAAE 50511415.1.0000.5546).

Trial design:

This study will be a randomized, triple-blind, placebo-controlled clinical trial with a cross-over design. The patients included will be submitted to two in-office bleaching sessions receiving placebo (control) or Piroxicam-beta-Cyclodextrin prior to the bleaching procedure; while different treatments will be allocated for each session. A delay of 1 week between the sessions (wash-out) will be established. The study will be conducted at the clinic of the School of Dentistry of the local university from December 2016 to May 2017.

Participants:

Patients included in this clinical trial will be at least 18 years old with good oral health. Patients with any of the six upper anterior teeth with caries lesions, restoration, severe discoloration (e.g., stains caused by tetracycline), fluorosis, gingival recession, dentin exposure, periodontal diseases, pulpitis, or endodontics treatment will be excluded. Participants submitted to previous bleaching procedures, presenting prior tooth sensitivity, known allergy to any component of medication used in the study, Continuous use of drugs with anti-inflammatory actions, pregnant or breastfeeding will be also excluded. Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (Vita Bleachguide 3D-Master scale, Vita-Zahnfabrik, Bad Sackingen, Germany) or darker will be included.

Sample Size Calculation:

The sample calculation will be based on the primary binary outcome (sensitivity risk 24 hours after the procedure) for superiority trial. Power of the test will be set at 80%, considering a type I error of 0.05; risk to tooth sensitivity of 90%, based on a prior study using similar bleaching agent, while a reduction around 30% with the treatment will be expected. The calculation resulted in fifty patients.

Randomization:

A randomized list will be computer-generated by a person not involved in intervention or evaluation. The participants were defined as blocks in the randomization process, where the sequence of treatment (placebo or piroxicam-beta-cyclodextrin) will be randomly set for each block by using computer-generated tables (www.sealedenvelope.com). The sequence will be inserted into sealed envelopes numbered from 1 to 50 that were opened by the operator only at the moment of the intervention. The patients were numbered according to the sequence of enrollment. Neither the participant nor the operator knew the group allocation determining blinding to the protocol.

Baseline evaluation:

Prior to bleaching procedure, the teeth will be cleaned using rubber cups associated to pumice and water. The shades of six upper anterior teeth will be assessed on a baseline using the bleach guide scale (Vita Bleach Guide,Vita-Zahnfabrik, Bad Säckinge, Germany). The shades' tabs selected will be converted to scores ranging from 1 (whiter shade - 0M1) to 15 (darker shade - 5M3).

Intervention:

Thirty minutes prior to each bleaching session, the patients will receive a capsule containing 20mg of piroxicam-beta-cyclodextrin or 20mg of placebo (inert content), according to the randomization, while the capsules will present the same appearance. The capsules with similar presentation will be manufactured by a person not involved in intervention or evaluation and will be placed into two bottles identified by letters according to treatment. Neither the operators responsible for intervention and evaluation nor the patients knew the content of each capsule.

A light-cured resin dam will be applied (Top Dam, FGM, Joinville, SC, Brazil) on the gingival tissue corresponding to the teeth to be bleached. A 35% hydrogen peroxide based bleaching agent (Whiteness HP Maxx, FGM, Joinville, SC, Brazil) will be mixed and applied on the vestibular surface of teeth, remaining for 45 minutes. After this time, the bleaching agent will be removed. A second session will beas carried out after 1 week following the same procedures. At this time, the patient received a single-dose capsule containing piroxicam-beta-cyclodextrin or placebo (different from the ones received at first session) thirty minutes before the procedure.

Evaluations:

The tooth sensitivity reported by patients will be recorded using both VAS and a verbal rating (VRS) scales. For VAS, the patient set her/his sensitivity level by pointing with a pen to the colored 10-cm scale and the distance from the border corresponding to absence of pain will be recorded. Tooth sensitivity will be also scored according to VRS, where 0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe.

The maximum level of tooth sensitivity will be evaluated during the bleaching procedure, during the first 24 hours and the level of sensitivity at that time. VRS will define the presence (score different from 0) or absence of tooth sensitivity in all time assessments. One week after each session the tooth color will be evaluated again using the same procedure described previously.

Statistical Analysis:

The demographic data from patients will be analyzed to determine age and gender for each allocation sequence. Comparisons between the allocation sequences will be performed by the Mann-Whitney test (age) and Fisher's exact (gender).

Based on presence of any tooth sensitivity (scores different from 0 for VRS), the absolute risk, odds ratio and relative risk will be calculated regarding the treatments for each moment of evaluation/session of bleaching, as well as its confidence intervals (95%). For each moment, differences on presence/absence ratios will be analyzed by Fisher's exact test. For the overall risk related to each treatment, the odds ratio will be adjusted to independent variable "session of bleaching" using the Mantel-Haenszel statistic. The homogeneity of odds ratios will be analyzed by the Breslow-Day and Tarone's tests. Following, the odds ratio estimated will be converted to relative risk and the overall presence/absence ratios will be analyzed by the McNemar's test, considering the study design (cross-over).

For VRS, the data from scores observed in each time of evaluation/session of bleaching will be submitted to the Mann-Whitney rank sum test. Despite the measurement of tooth sensitivity using VAS giving a continuous outcome, data assessed with this scale did not show a normal distribution (Shapiro-Wilk's test). Thus, data from VAS will be also analyzed by the Mann-Whitney rank sum test, while one test per time of evaluation will be carried out.

For color evaluation, comparisons between the sequences of treatment will be performed using the Mann-Whitney rank sum test. The Friedman test followed by Dunn's post hoc test will be used to analyze the difference between the moments of evaluation for each sequence of treatment. All statistical analyses will be performed adjusting the initial significance level (α = 0.05) by Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old patients of both genders presenting good general/oral health;
* All maxillary anterior teeth presenting shade equal or darker than 2,5M2 at Vita bleachguide guide (Vita-Zahnfabrik, Germany);
* Signed the form accepting to participate of this study.

Exclusion Criteria:

* Presence of caries lesions, restorations and/or endodontic treatment at any maxillary anterior teeth.
* Undergone tooth-whitening procedures;
* Pregnant/lactating;
* Presence of periodontal diseases;
* Presence of severe tooth discoloration by tetracycline stains or fluorosis;
* Any kind of medicine, bruxism habits or any other pathology that can cause sensitivity (such as recession, dentin exposure);
* Continuous use of drugs with anti-inflammatory actions;
* Presence of tooth hypersensitivity at baseline measurement;
* Any known adverse effects caused by Piroxicam-beta-Cyclodextrin;
* Non-attendance to any session of evaluation or bleaching.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Risk to Tooth sensitivity | up to 24 hours after each session. [Safety Issue: Yes]
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Level to Tooth sensitivity | up to 24 hours after each session.[Safety Issue: Yes
  The tooth sensitivity also will be evaluated using a analogic visual analogue (VAS) consisted of a scale 10 cm in length ranging from 0 (absence of pain) to 10 (unsupportable pain). The patient set his or her level of sensitivity by pointing on the scale corresponding to this level, while the distance from this point to the 0 border will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aline C Peixoto, Principal Investigator — Universidade Federal de Sergipe
Locations (1):
- Hospital Universitário - Universidade Federal de Sergipe, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: No